CLINICAL TRIAL: NCT01908062
Title: Comparing Treatments for HIV-Infected Opioid and Alcohol Users in an Integrated Care Effectiveness Study
Acronym: CHOICES
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, P. Todd Korthuis, MD, Associate Professor of Medicine, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIDA-CTN-0055; U10DA015815 (NIH)
Record Dates: First submitted 2013-07-23; First posted 2013-07-25 (Estimated); Results first posted 2019-02-26 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Opioid Use Disorder; Alcohol Use Disorder
Keywords: Substance related disorders; HIV; naltrexone
MeSH Terms: conditions — Opioid-Related Disorders; Alcoholism; Substance-Related Disorders | interventions — vivitrol; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment as Usual (Active Comparator): The current standard of care for treatment of opioid use disorders in HIV clinics is opioid agonist therapy. HIV-infected patients with alcohol use disorders are typically referred for residential, outpatient, and self-help groups.
  Interventions: Other: Treatment As usual
- Extended Release Naltrexone (Experimental): Extended release naltrexone (XR-NTX), delivered by monthly injection. Dose: 380 mg. Frequency: One injection per month, for four months. Duration: 30 days.
  Interventions: Drug: Extended Release Naltrexone

INTERVENTIONS:
Drug: Extended Release Naltrexone
  Other Names: Vivitrol
  Arms: Extended Release Naltrexone
Other: Treatment As usual
  Arms: Treatment as Usual

SUMMARY:
The purpose of this study is to learn how best to treat substance use disorders in an HIV clinic setting. Specifically, the purpose of this pilot study is to learn if extended-release naltrexone (XR-NTX) would be a feasible and acceptable treatment for HIV-infected individuals with opioid or alcohol use disorders.

ELIGIBILITY:
Inclusion Criteria:

1. Meet Diagnostic and Statistical Manual (DSM-5) criteria for moderate or severe opioid use disorder and/or alcohol use disorder.
2. Be willing to be randomized to antagonist-based therapy or treatment as usual (TAU) for treatment of opioid and/or alcohol use disorders.
3. Be HIV-infected as defined by history of positive HIV serology or HIV RNA pcr >10,000 copies/mL).
4. Be willing to establish ongoing HIV care at community treatment program(CTP) if not already receiving ongoing care.
5. Be willing to initiate antiretroviral therapy (ART) if not already prescribed ART, regardless of CD4 count.
6. Be at least 18 years old.
7. Be able to provide written informed consent and HIPAA (if applicable) for medical record abstraction.
8. Be able to communicate in English.
9. If female, be willing to take measures to avoid becoming pregnant.

Exclusion Criteria:

Individuals will be excluded from pilot study participation if they:

* Have a serious medical, psychiatric or substance use disorder that, in the opinion of the study physician, would make study participation hazardous to the participant, compromise study findings, or prevent the participant from completing the study.

Examples include:

1. Disabling or terminal medical illness (e.g., active opportunistic infection, uncompensated heart failure, cirrhosis or end-stage liver disease, acute hepatitis and moderate to severe renal impairment) as assessed by medical history, review of systems, physical exam and/or laboratory assessments;

   1. Severe, untreated or inadequately treated mental health disorder (e.g., active psychosis, uncontrolled manic-depressive illness) as assessed by history and/or clinical interview;
   2. Current severe benzodiazepine or other depressant or sedative hypnotic use requiring medical detoxification;
   3. Suicidal or homicidal ideation requiring immediate attention.
2. Have aspartate aminotransferase (AST) or alanine aminotransferase (ALT) liver enzymes greater than 5 times upper limit of normal on screening phlebotomy. Results from tests conducted within the past 30 days which are abstracted from medical record information are acceptable.
3. Have international normalized ratio (INR) > 1.5 or platelet count <100k. Results from tests conducted within the past 30 days which are abstracted from medical record information are acceptable.
4. Have known allergy or sensitivity to naloxone, naltrexone, polylactide-co-glycolide, carboxymethylcellulose, or other components of the Vivitrol® diluents.
5. Anticipate undergoing surgery during study participation.
6. Have chronic pain requiring ongoing pain management with opioid analgesics.
7. Pending legal action or other reasons that might prevent an individual from completing the study.
8. Currently pregnant or breastfeeding.
9. Body habitus that, in the judgment of the study physician, precludes safe intramuscular injection of XR-NTX, (e.g. excess fat tissue over the buttocks).
10. Received methadone or buprenorphine maintenance therapy for treatment of opioid dependence in the 4 weeks prior to screening.
11. Have taken an investigational drug in another study within 30 days of study consent.
12. Have ECG findings that, in the opinion of the study medical clinician would preclude safe participation in the study. Results from ECGs conducted within the past 30 days which are abstracted from medical record information are acceptable.
13. Have had treatment with XR-NTX for opioid or alcohol dependence in the 3 months prior to screening.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2014-06; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip T Korthuis, MD, MPH, Principal Investigator — Oregon Health and Science University
Locations (2):
- The CORE Center, Chicago, Illinois, United States
- University of British Columbia, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Kornor H, Lobmaier PPK, Kunoe N. Sustained-release naltrexone for opioid dependence. Cochrane Database Syst Rev. 2025 May 9;5(5):CD006140. doi: 10.1002/14651858.CD006140.pub3. PMID 40342086
- [Derived] Korthuis PT, Lum PJ, Vergara-Rodriguez P, Ahamad K, Wood E, Kunkel LE, Oden NL, Lindblad R, Sorensen JL, Arenas V, Ha D, Mandler RN, McCarty D; CTN-0055 CHOICES Investigators. Feasibility and safety of extended-release naltrexone treatment of opioid and alcohol use disorder in HIV clinics: a pilot/feasibility randomized trial. Addiction. 2017 Jun;112(6):1036-1044. doi: 10.1111/add.13753. Epub 2017 Feb 8. PMID 28061017

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment as Usual: The current standard of care for treatment of opioid use disorders in HIV clinics is opioid agonist therapy. HIV-infected patients with alcohol use disorders are typically referred for residential, outpatient, and self-help groups.
  Treatment As usual
- Extended Release Naltrexone: Extended release naltrexone (XR-NTX), delivered by monthly injection. Dose: 380 mg. Frequency: One injection per month, for four months. Duration: 30 days.
  Extended Release Naltrexone
Period: Overall Study
Arm/Group | Treatment as Usual | Extended Release Naltrexone
Started | 26 | 25
Completed | 24 | 22
Not Completed | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment as Usual | Extended Release Naltrexone | Total
Number analyzed (Participants) | 26 | 25 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (12) | 47 (8.8) | 46 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 14 | 22
  Male | 18 | 11 | 29
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 12 | 12 | 24
  United States | 14 | 13 | 27

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Successful Initiation of Treatment Within 4 Weeks of Randomization
Description: Successful induction onto XR-NTX or initiation of treatment as usual within 4 weeks of randomization.
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment as Usual | Extended Release Naltrexone
Number analyzed (Participants) | 26 | 25
Participants | 25 | 17

2. Primary Outcome: Number of Participants Successfully Retained on Pharmacotherapy Treatment at 16 Weeks
Description: Number of participants who received the maximum possible expected doses of XR-NTX, or the full course of recommended pharmacotherapy treatment for treatment as usual (TAU) arm.
Time Frame: 16 weeks
Population: 24 TAU participants, and 17 XR-NTX participants initiated treatment in their respective arms. Treatment retention is calculated only for subjects who have been initiated onto treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Treatment as Usual Pharmacotherapy: The current standard of care for treatment of opioid use disorders in HIV clinics is opioid agonist therapy. Pharmacotherapy for TAU participants with alcohol use disorder (AUD) consisted of oral naltrexone, gabapentin, acamprosate, and disulfiram.
  Treatment As usual
Arm/Group | Treatment as Usual Pharmacotherapy | Extended Release Naltrexone
Number analyzed (Participants) | 24 | 17
Participants | 12 | 15

3. Secondary Outcome: HIV Viral Suppression at 16 Weeks
Description: Plasma HIV viral load of < 200 copies/mL compared with screening
Time Frame: 16 weeks
Population: 23 TAU participants and 21 XR-NTX participants had a 16-week lab draw for HIV viral load testing.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment as Usual | Extended Release Naltrexone
Number analyzed (Participants) | 23 | 21
Participants | 20 | 17

4. Secondary Outcome: Mean Days of Opioid Use in Past 30 Days
Description: Change in 30 day opioid use by Addiction Severity Index (ASI)-lite self-report and Time-Line Follow Back in the final 30 days of the 16 week trial compared to screening.
Time Frame: Baseline and 16 weeks
Population: In both the TAU and XR-NTX groups, reporting results for participants who were retained at 16 weeks and completed necessary study assessments.
Measure: Mean (Standard Deviation); unit: days
Groups:
- Treatment as Usual: The current standard of care for treatment of opioid use disorders in HIV clinics is opioid agonist therapy.
  Treatment As usual
Arm/Group | Treatment as Usual | Extended Release Naltrexone
Number analyzed (Participants) | 12 | 12
days
  Baseline mean days opioid use in past 30 days | 17.3 (13.14) | 20.3 (12.29)
  16 weeks mean days opioid use in past 30 days: number analyzed (Participants) | 11 | 11
  16 weeks mean days opioid use in past 30 days | 4.1 (5.43) | 7.7 (11.32)

5. Secondary Outcome: HIV Care Engagement
Description: Change in the proportion of participants prescribed antiretroviral therapy (ART) within 16 weeks following randomization, compared to baseline.
Time Frame: Baseline and 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment as Usual | Extended Release Naltrexone
Number analyzed (Participants) | 26 | 25
Participants
  Prescribed ART at baseline | 25 | 23
  Prescribed ART at 16 weeks | 26 | 24

6. Secondary Outcome: Participant Safety: Change in Liver Enzymes Between Baseline and Week 16
Description: Change in liver enzymes between screening and Week 16. AST = Aspartate transaminase ALT = Alanine transaminase
Time Frame: Baseline and 16 weeks
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Treatment as Usual | Extended Release Naltrexone
Number analyzed (Participants) | 26 | 25
IU/L
  Mean AST at baseline | 32.3 (19.4) | 36.8 (23.1)
  Mean AST at 16 weeks | 32.2 (17.6) | 38.8 (27.6)
  Mean ALT at baseline | 33.0 (24.5) | 35.0 (35.6)
  Mean ALT at 16 weeks | 30.8 (18.1) | 40.1 (38.4)

7. Secondary Outcome: Number of Participants With Urine Drug Screen (UDS) Positive for Opioids
Time Frame: Baseline and 16 weeks
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment as Usual | Extended Release Naltrexone
Number analyzed (Participants) | 12 | 12
Participants
  Baseline UDS positive for opioids | 9 | 9
  16 weeks UDS positive for opioids | 7 | 4

8. Secondary Outcome: Mean Days of Alcohol Use in Past 30 Days
Description: Change in 30 day alcohol use by Addiction Severity Index (ASI)-lite self-report and Time-Line Follow Back in the final 30 days of the 16 week trial compared to screening.
Time Frame: Baseline and 16 weeks
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Treatment as Usual | Extended Release Naltrexone
Number analyzed (Participants) | 14 | 13
days
  Baseline mean days alcohol use in past 30 days | 15.6 (9.95) | 12.5 (11.02)
  16 weeks mean days alcohol use in past 30 days | 5.7 (8.40) | 2.8 (3.05)

9. Secondary Outcome: Number of Participants With Urine Ethyl Glucuronide (EtG) Positive for Alcohol
Time Frame: Baseline and 16 weeks
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment as Usual | Extended Release Naltrexone
Number analyzed (Participants) | 14 | 13
Participants
  Baseline EtG positive for alcohol | 7 | 6
  16 weeks EtG positive for alcohol | 4 | 3

10. Secondary Outcome: Participant Safety: Any Fatal or Non-fatal Overdose Between Baseline and Week 16
Time Frame: 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment as Usual | Extended Release Naltrexone
Number analyzed (Participants) | 26 | 25
Participants
  Nonfatal opioid overdose | 1 | 1
  Fatal opioid overdose | 0 | 0

11. Secondary Outcome: Participant Safety: Precipitated Withdrawal
Description: Proportion of participants assigned to XR-NTX who develop precipitated opioid withdrawal.
Time Frame: 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Extended Release Naltrexone
Number analyzed (Participants) | 25
Participants | 0

ADVERSE EVENTS:
Arm/Group | Treatment as Usual | Extended Release Naltrexone
Serious Adverse Events (participants affected / at risk) | 1/26 | 1/25
Other Adverse Events (participants affected / at risk) | 5/26 | 9/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment as Usual (N=26) | Extended Release Naltrexone (N=25)
Suicidal Ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Ankle Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment as Usual (N=26) | Extended Release Naltrexone (N=25)
Diarrhea (Gastrointestinal disorders) | 0 | 2
Headache, Migraine (Nervous system disorders) | 1 (26) | 2 (25)
Nausea (Gastrointestinal disorders) | 4 | 4
Vomiting (Gastrointestinal disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No